CLINICAL TRIAL: NCT06941025
Title: Maternal and Postnatal Outcomes Study (MOS) A Worldwide Decentralized Observational Registry to Evaluate the Safety in Women With Fabry Disease and Their Infants Exposed to Elfabrio® (Pegunigalsidase Alfa-iwxj/Pegunigalsidase Alfa) During Pregnancy and/or Lactation
Brief Title: Maternal and Postnatal Outcomes Study (MOS): A Global Observational Registry Assessing the Safety of Elfabrio® in Women With Fabry Disease and Their Infants During Pregnancy and Breastfeeding
Acronym: MOS
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-06657AA1-06
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Fabry Disease; Pregnancy; Pregnancy Complications
MeSH Terms: conditions — Fabry Disease; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Fabry disease who were exposed to pegunigalsidase alfa during pregnancy and/or lactation
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable - observational study

SUMMARY:
The goal of this observational registry is to evaluate the safety and outcomes of pregnancy and lactation in women with Fabry disease who are exposed to pegunigalsidase alfa within 30 days prior to conception and/or during pregnancy and lactation.

The main objectives are to:

* Assess pregnancy outcomes, including maternal and infant health.
* Evaluate the occurrence of congenital malformations and other neonatal outcomes.

This is a global, decentralized, single-arm, prospective and retrospective registry planned to enroll participants over a 10-year period. Eligible patients may be enrolled by their physician or may self-enroll, where permitted by local regulations. Data will be collected through a secure web-based platform, allowing patients and physicians to enter information via electronic case report forms (eCRFs).

Pregnancy and clinical outcomes will be documented throughout pregnancy and up to 12 months post-birth. Data from self-enrolled patients will be confirmed by their primary care or attending physician. This registry is observational and does not impact clinical care or treatment decisions.

DETAILED DESCRIPTION:
This is a global, decentralized, single-arm, prospective and retrospective observational registry designed to evaluate pregnancy and infant outcomes in women with Fabry disease who have been exposed to pegunigalsidase alfa within 30 days prior to conception and/or during pregnancy and lactation. The registry aims to assess maternal and infant safety, pregnancy outcomes, and the occurrence of congenital malformations and other neonatal conditions.

The registry will enroll patients over a 10-year period. Eligible patients may be enrolled by their physician or may self-enroll, where permitted by local regulations. Data collection will be facilitated through a secure, centralized web-based platform, where patients and physicians can enter information using electronic case report forms (eCRFs).

Enrollment & Data Collection:

Patients can be enrolled at any time, either during pregnancy or after delivery. Depending on the timing of enrollment, data will be collected retrospectively and/or prospectively.

Pregnancy and clinical outcomes will be monitored from enrollment until the infant reaches 12 months of age.

Collected data includes maternal health, pregnancy complications, delivery outcomes, congenital malformations, and infant health parameters.

Reported congenital malformations will be classified according to established criteria (e.g., MACDP, EUROCAT) and adjudicated by an independent Scientific Advisory Committee.

The registry is observational and does not alter clinical care, physician treatment decisions, or patient management.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with Fabry disease who have been exposed to at least 1 dose of pegunigalsidase alfa at any time during pregnancy (defined as having received pegunigalsidase alfa within 30 days prior to the DOC and/or during pregnancy) and/or during lactation, and their infants.

  o DOC, defined as 20/7 gestational weeks, will be calculated from last menstrual period [LMP] or ultrasound
* Patient or parent/legally authorized representative must be able to understand and provide consent through an Institutional Review Board / Independent Ethics Committee (IRB/IEC) approved Informed Consent Form.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant and/or breastfeeding women with Fabry disease and their infants, after exposure to at least 1 dose of pegunigalsidase alfa during pregnancy and/or during lactation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcome: Number of live births | at the delivery, after an average of 40 weeks of pregnancy
Pregnancy outcome: Number of preterm birth | at delivery, prior to 37 weeks of gestation
Pregnancy outcome: Number of pregnancy losses (number of spontaneous abortions , number of pregnancy terminations, number of foetal deaths or stillbirths) | spontaneous abortions: up to 20 weeks of pregnancy; pregnancy terminations: through the pregnancy; number of foetal deaths or stillbirths: greater than 20 weeks of pregnancy and through the pregnancy, average of 40 weeks

SECONDARY OUTCOMES:
Number of neonates/infants with MCMs | through the pregnancy, an average of 40 weeks and up to 12 months of infant age
Number of ectopic or molar pregnancies | through the pregnancy, an average of 40 weeks
Number of women with obstetric and delivery complications | at the delivery, an average of 40 weeks of pregnancy
Number of women with complications of preeclampsia or eclampsia | through the pregnancy, an average of 40 weeks
Number of women with complications of preterm prelabour rupture of membrane | at delivery, prior to 37 weeks of gestation
Number of neonates/infants with minor congenital malformations | through the pregnancy, an average of 40 weeks and up to 12 months of infant age
Number of infants with developmental deficiency | up to 12 months of infant age
Number of hospitalisations in infants | up to 12 months of infant age
Mortality in infants, including neonatal death and infant death | up to 12 months of infant age
Head circumference in infants (cm) | up to 12 months of infant age
Weight in infants (kilograms) | up to 12 months of infant age
Length in infants (cm) | up to 12 months of infant age
Number of infants born as SGA | up to 12 months of infant age
Number of infants with postnatal growth deficiency or FTT | up to 12 months of infant age
Duration of breastfeeding, number of exclusively breastfeeding women and number of breastfeeding women supplemented with formula | up to 12 months of infant age
Number of adverse events in infants exposed to pegunigalsidase alfa during breastfeeding | up to 12 months of infant age

CONTACTS AND LOCATIONS:
Locations (5):
- No physical study sites - Decentralized, web-based registry, Washington D.C., District of Columbia, United States
- No physical study sites - Decentralized, web-based registry, Berlin, Germany
- No physical study sites - Decentralized, web-based registry, Rome, Italy
- No physical study sites - Decentralized, web-based registry, Madrid, Spain
- No physical study sites - Decentralized, web-based registry, London, United Kingdom

REFERENCES:
- See also: Official registry website with information on eligibility, participation, and data collection for the observational study on pregnancy and infant outcomes in women with Fabry disease. — https://elfabriopregnancyregistry.com
- See also: Official registry website with information on eligibility, participation, and data collection for the observational study on pregnancy and infant outcomes in women with Fabry disease. — https://mospregnancyregistry.com